CLINICAL TRIAL: NCT04802031
Title: Safety of Rapid-Infusion Isatuximab in Patients With Relapsed/Refractory Multiple Myeloma
Brief Title: Rapid-infusion Isatuximab in Relapsed/Refractory Multiple Myeloma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual
Sponsor: Thomas Martin, MD (Other)
Responsible Party: Sponsor-Investigator, Thomas Martin, MD, Principal Investigator, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202530; NCI-2021-01226 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2021-03-13; First posted 2021-03-17 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Relapsed Multiple Myeloma; Refractory Multiple Myeloma
Keywords: Isatuximab Infusion
MeSH Terms: conditions — Multiple Myeloma | interventions — isatuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (isatuximab) (Experimental): Participants receive their first rapid infusion of isatuximab IV over 30 minutes. If a >=Grade 2 iRR occurs, then participants will revert to a SOC infusion time and be removed from the study. If a Grade 1 or no IRR occurs, then participants will receive another rapid infusion of 30 minutes. Participants will continue to receive RI and IRR assessment after each dose up to at least 6 doses or until a grade 2 or higher IRR occurs.
  Interventions: Biological: Rapid Infusion Isatuximab

INTERVENTIONS:
Biological: Rapid Infusion Isatuximab — Given IV
  Other Names: Hu 38SB19; ISATUXIMAB; Isatuximab-irfc; SAR 650984; SAR650984; Sarclisa

SUMMARY:
This phase II trial studies the effects of isatuximab given as a rapid-infusion in treating multiple myeloma that has come back (recurrent) or has not responded to treatment (refractory). Isatuximab, also known as Sarclisa, is an antibody (proteins that can protect the body from foreign organisms, such as bacteria and viruses) directed against cluster of differentiation 38 (CD38), a receptor antigen (a receptor or protein on the outside of blood cells that can be used as a target). Isatuximab may stop the growth of some blood cancers. Normally, the fastest that intravenous isatuximab can be given - for patients who have not had any reactions to their first two doses - is over 1 hour and 15 minutes. This study is designed to test whether intravenous isatuximab can be given over 30 minutes ("rapid infusion") among patients who have not developed any reactions to at least 2 prior doses of intravenous isatuximab at normal speeds. If shown to be safe, "rapid infusion" isatuximab may ultimately improve the patient experience while reducing the overall cost of the infusion.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the incidence of grade 2 or higher (Gr2+) infusion-related reactions (IRRs) with rapid-infusion (RI) isatuximab across 6 doses.

SECONDARY OBJECTIVE:

I. To estimate time savings with RI isatuximab (versus estimated standard of care [SOC] isatuximab duration lengths) across 6 doses of isatuximab.

OUTLINE:

Patients must have received standard of care isatuximab IV over for at least 2 doses without any Gr2+ IRRs reported. Patients will then receive a rapid infusion of isatuximab IV over 30 minutes. If a >=Grade 2 iRR occurs, then participants will revert to a SOC infusion time and be taken off the study. If a Grade 1 or no IRR occurs, then participants will receive another rapid infusion of 30 minutes and assessed again for IRRs. Rapid infusions and IRR assessment after each RI will continue for up to at least 6 doses or until the patient experiences an Grade 2 or higher IRR.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of multiple myeloma (International Classification of Disease (ICD-10) code: C90.0)
* Previous exposure to at least one proteasome inhibitors (PI) and lenalidomide (or candidacy for isatuximab as per updated Food and Drug Administration (FDA) package insert information in the future)
* Planned or current isatuximab-containing therapy. Patients receiving isatuximab as part of a clinical trial are eligible for this study if allowed by the trial sponsor.

  * For ease of registration, patients will be allowed to enroll at any point after the decision is made to initiate isatuximab (with the understanding that their initial doses will be standard of care (SOC), including the first 2 doses for all patients). However, rapid infusion (RI) isatuximab will only be administered to participants who have not had infusion-related reactions (iRRs) during >= 2 consecutive prior doses of SOC isatuximab
* Ability to understand a written informed consent form (ICF) document, and the willingness to sign the ICF document

Exclusion Criteria:

* Age < 18
* Body weight > 70 kilograms (kg) at the time of any RI isatuximab dose
* Current pregnancy or (if of reproductive age) unwillingness to follow contraception requirements as per the FDA package insert
* New York Heart Association Stage IV heart disease, i.e. unable to carry on any physical activity without discomfort or symptoms of heart failure (as per study investigator)
* Any medical condition, including mental illness or substance abuse, deemed by the principal investigator to interfere with the ability to provide consent or cooperate with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-05-28 (Actual); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with reported grade 2 or higher infusion-related reactions (IRR) | Up to 6 months
  The per-patient incidence of Grade 2 or higher IRRs with rapid infusion (RI) isatuximab will be calculated as the number of patients who developed >= 1 Grade 2+ IRR with RI isatuximab divided by the total number of patients who receive >= 1 dose of RI isatuximab.

SECONDARY OUTCOMES:
Mean per-participant infusion duration | 9-12 weeks depending on isatuximab dosing interval
  Descriptive statistics for total infusion durations in minutes including mean, standard deviation, and 95% confidence interval will be reported across the first 6 doses of RI isatuximab.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Martin, MD, Principal Investigator — University of California, San Francisco

IPD SHARING:
Plan to Share IPD: No